CLINICAL TRIAL: NCT04374851
Title: A Comparative Clinical Investigation of Two Hearing Instrument Digital Signal Processing Strategies and Their Effect on Speech Understanding
Brief Title: A Comparative Clinical Investigation of Two Hearing Instrument Digital Signal Processing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bernafon AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: BF005-2000
Record Dates: First submitted 2020-04-16; First posted 2020-05-05 (Actual); Last update posted 2021-01-07 (Actual); Status verified 2021-01

CONDITIONS: Hearing Loss
MeSH Terms: conditions — Hearing Loss

STUDY DESIGN:
Intervention Model Description: Subjects will randomly wear the new device or the current device for the first period and then switch to the other device for the second period.
Who Masked: Participant, Investigator
Masking Description: The subjects will not know which device they are using in each period (new or current) because they look exactly the same. The PI will also not know which device is used as they will be prepared for the PI before the Appointments.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- New Device (Experimental): The new Hearing aid is essentially the same as the current device (i.e., hardware, use) but with an improved digital signal processing (DSP).
  Interventions: Device: Polaris miniRITE BTE
- Current Device (Active Comparator): The current device is the Hearing aid that is currently sold on the market. It is used as a normal Hearing aid that is worn daily to amplify sounds for Hearing-impaired people.
  Interventions: Device: Viron miniRiTE BTE

INTERVENTIONS:
Device: Polaris miniRITE BTE — The Polaris device is programmed with computer software to match the Hearing loss of the participant.
  Arms: New Device
Device: Viron miniRiTE BTE — The Viron Hearing device is programmed with computer software to match the Hearing loss of the participant.
  Arms: Current Device

SUMMARY:
The purpose of this study is to show that the performance of the new digital signal processing system is better than the system used in the currently CE marked devices. Speech in narrowband noise and acceptable levels of noise should be improved with the new system, and speech understanding overall should not be negatively affected. There should be no artefacts or unwanted noises caused by the new system.

DETAILED DESCRIPTION:
This is a controlled, double-blinded, comparative clinical evaluation conducted monocentric at the premised of Bernafon AG in Bern, Switzerland.

For this study, Bernafon AG will carry out testing with participants with hearing loss to validate the performance of a new digital signal processing (DSP). System testing of the DSP shows an improved signal, yet it must be tested with humans to be sure of an improvement in real-life situations. The current study will compare the new DSP to the one that is used in the Bernafon hearing aids that are CE- marked and currently available on the market. The goal is to determine whether the new DSP is better in real-life situations than the current system.

Primary Endpoint: The primary objective is to assess the new DSP system with various hearing losses and levels of amplification. Speech testing will be used to analyse the speech perception of participants.

Secondary Endpoint: The secondary objective is to verify the overall performance of the new device. Acceptable noise levels will be measured as well as further speech testing. Questionnaires will be used to measure subjective responses to the performance.

Other Endpoints: The subjective performance of an optimized fitting versus a standard fitting and the acceptance of new domes will be measured with questionnaires.

Safety Endpoint: The study aims to identify any new risk factors and to ensure the safety of the device with the newly implemented DSP system before releasing it to the market.

ELIGIBILITY:
Inclusion Criteria:

* Hearing loss (sensorineural, conductive, mixed-must have doctor approval for mixed and conductive Hearing loss)
* Severity of Hearing loss ranging from mild to profound
* German speaking
* Current Hearing aid users
* Ability and willingness to sign the consent form

Exclusion Criteria:

* Contraindications for amplification
* New Hearing aid users
* Inability to follow the procedures
* Inability to attend Weekly study Appointments
* Strongly reduced dexterity
* Central Hearing disorders
* Bernafon employees
* Family members of Bernafon employees

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2020-08-03 (Actual); Primary Completion 2020-11-30 (Actual); Study Completion 2020-11-30 (Actual)

PRIMARY OUTCOMES:
Speech perception with narrowband noise | Week 1
  Speech perception is tested using a standardized speech test that requires subjects to repeat sentences presented among narrowband background noise. The test is adaptive with the background noise getting louder or softer so that the subject answers 50% correct. The scores are measured in dB SNR (signal-to-noise ratio) and a lower score is better. The lowest possible score is -15 dB SNR and the highest is +20 dB SNR. It is measured in the unaided condition.
Speech perception with narrowband noise | Week 2
  Speech perception is tested using a standardized speech test that requires subjects to repeat sentences presented among narrowband background noise. The test is adaptive with the background noise getting louder or softer so that the subject answers 50% correct. The scores are measured in dB SNR (signal-to-noise ratio) and a lower score is better. The lowest possible score is -15 dB SNR and the highest is +20 dB SNR. It is measured in the aided condition with the new device or the current device depending on the randomization.
Speech perception with narrowband noise | Week 3
  Speech perception is tested using a standardized speech test that requires subjects to repeat sentences presented among narrowband background noise. The test is adaptive with the background noise getting louder or softer so that the subject answers 50% correct. The scores are measured in dB SNR (signal-to-noise ratio) and a lower score is better. The lowest possible score is -15 dB SNR and the highest is +20 dB SNR. It is measured in the aided condition with the new device or the current device depending on the randomization.

SECONDARY OUTCOMES:
Speech perception with broadband noise | Week 1
  Speech perception is tested using a standardized speech test that requires subjects to repeat sentences presented among broadband background noise. The test is adaptive with the background noise getting louder or softer so that the subject answers 50% correct. The scores are measured in dB SNR (signal-to-noise ratio) and a lower score is better. The lowest possible score is -15 dB SNR and the highest is +20 dB SNR. It is measured in the unaided condition.
Speech perception with broadband noise | Week 2
  Speech perception is tested using a standardized speech test that requires subjects to repeat sentences presented among broadband background noise. The test is adaptive with the background noise getting louder or softer so that the subject answers 50% correct. The scores are measured in dB SNR (signal-to-noise ratio) and a lower score is better. The lowest possible score is -15 dB SNR and the highest is +20 dB SNR. It is measured in the aided condition with the new device or the current device depending on the randomization.
Speech perception with broadband noise | Week 3
  Speech perception is tested using a standardized speech test that requires subjects to repeat sentences presented among broadband background noise. The test is adaptive with the background noise getting louder or softer so that the subject answers 50% correct. The scores are measured in dB SNR (signal-to-noise ratio) and a lower score is better. The lowest possible score is -15 dB SNR and the highest is +20 dB SNR. It is measured in the aided condition with the new device or the current device depending on the randomization.
Acceptance of noise | Week 1
  Acceptance of noise is tested using a standardized noise test that requires the subjects to adjust the background noise to the maximum Levels that they can tolerate it and to the Levels at which they can understand speech. It is measured in dB SNR (signal-to-noise ratio) and a lower score is better. The lowest score possible is -25 dB SNR and the highest is +20 dB SNR. It is measured in the unaided condition.
Acceptance of noise | Week 2
  Acceptance of noise is tested using a standardized noise test that requires the subjects to adjust the background noise to the maximum Levels that they can tolerate it and to the Levels at which they can understand speech. It is measured in dB SNR (signal-to-noise ratio) and a lower score is better. The lowest score possible is -25 dB SNR and the highest is +20 dB SNR. It is measured in the aided condition with the new device or the current device depending on the randomization.
Acceptance of noise | Week 3
  Acceptance of noise is tested using a standardized noise test that requires the subjects to adjust the background noise to the maximum Levels that they can tolerate it and to the Levels at which they can understand speech. It is measured in dB SNR (signal-to-noise ratio) and a lower score is better. The lowest score possible is -25 dB SNR and the highest is +20 dB SNR. It is measured in the aided condition with the new device or the current device depending on the randomization.

OTHER OUTCOMES:
Preference for Standard or Optimized Fitting | Week 5
  The Hearing aids will be programmed with a standard or default Fitting from the software and with an optimized Fitting based on questions answered by the subjects. At the end of a field test using both Fittings they will answer a questionnaire asking them to choose a preferred Fitting. They will have a scale from 1 to 10 to say how sure they are about their choice (1 being unsure and 10 being completely sure). They will also choose from a list of options reasons for giving their choice (i.e., speech intelligibility, Sound Quality, feedback).

CONTACTS AND LOCATIONS:
Overall Officials: Barbara Simon, AuD, Principal Investigator — Bernafon AG
Locations (1):
- Bernafon AG, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: No
There is no plan to share individual data.